CLINICAL TRIAL: NCT00714961
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Comparing Clopidogrel Plus Acetylsalicylic Acid (ASA) Versus ASA Alone in Subjects With Acute ST Elevation Myocardial Infarction (STEMI) Treated With Fibrinolytic Therapy
Brief Title: Clopidogrel as Adjunctive Reperfusion Therapy - Thrombolysis in Myocardial Infarction
Acronym: CLARITY-TIMI28
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EFC5133; CV149-015
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Clopidogrel (SR25990)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clopidogrel (SR25990) — plus acetylsalicylic acid (ASA)
  Arms: 1
Drug: Placebo — plus acetylsalicylic acid (ASA)
  Arms: 2

SUMMARY:
The purpose of this study is to determine if the combination of aspirin plus clopidogrel is more effective than aspirin alone in preventing another heart attack, chest pain, stroke or death in people who have already had a heart attack that was treated with fibrinolytic therapy.

ELIGIBILITY:
Inclusion Criteria:

* STEMI within 12 hours of randomization
* Planned treatment with a fibrinolytic agent and aspirin

Exclusion Criteria:

* Intention of performing coronary angiography within 48 hours of fibrinolysis
* Treatment with clopidogrel or ticlopidine within 7 days prior to enrollment, or planned treatment with clopidogrel or ticlopidine.
* Contraindication to fibrinolysis
* Planned use of a glycoprotein IIb/IIIa inhibitor
* Prior CABG
* Evidence of cardiogenic shock or acute pulmonary edema requiring intubation or an intraaortic balloon pump
* Known renal or hepatic insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3491 (Actual)
Dates: Start 2003-02; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
efficacy: composite of an included infarct-related artery on the pre-discharge angiogram, or death or recurrent MI by the time of the start of coronary angiography
safety: TIMI major bleeding

SECONDARY OUTCOMES:
Angiographic, clinical and electrocardiographic outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Braunwald, MD, Principal Investigator — Brigham and Women's Hospital, Boston, MA, USA
Locations (24):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Buenos Aires, Argentina
- Sanofi-Aventis, Macquarie Park, Australia
- sanofi-aventis Austria, Vienna, Austria
- sanofi-aventis Belgium, Diegem, Belgium
- sanofi-aventis Brazil, São Paulo, Brazil
- sanofi-aventis Canada, Laval, Canada
- sanofi-aventis France, Paris, France
- sanofi-aventis Germany, Berlin, Germany
- Sanofi-Aventis Hungaria, Budapest, Hungary
- Sanofi-Aventis, Dublin, Ireland
- Sanofi-Aventis, Netanya, Israel
- sanofi-aventis Italy, Milan, Italy
- Sanofi-Aventis Mexico, México, Mexico
- sanofi-aventis Netherlands, Gouda, Netherlands
- sanofi-aventis Poland, Warsaw, Poland
- Sanofi-Aventis, Porto, Portugal
- Sanofi-Aventis, San Juan, Puerto Rico
- Sanofi-Aventis, Moscow, Russia
- sanofi-aventis South Africa, Midrand, South Africa
- sanofi-aventis Spain, Barcelona, Spain
- sanofi-aventis Sweden, Bromma, Sweden
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)
- sanofi-aventis UK, Guildford, United Kingdom

REFERENCES:
- [Result] Sabatine MS, Cannon CP, Gibson CM, Lopez-Sendon JL, Montalescot G, Theroux P, Claeys MJ, Cools F, Hill KA, Skene AM, McCabe CH, Braunwald E; CLARITY-TIMI 28 Investigators. Addition of clopidogrel to aspirin and fibrinolytic therapy for myocardial infarction with ST-segment elevation. N Engl J Med. 2005 Mar 24;352(12):1179-89. doi: 10.1056/NEJMoa050522. Epub 2005 Mar 9. PMID 15758000
- [Derived] Harkness JR, Sabatine MS, Braunwald E, Morrow DA, Sloan S, Wiviott SD, Giugliano RP, Antman EM, Cannon CP, Scirica BM. Extent of ST-segment resolution after fibrinolysis adds improved risk stratification to clinical risk score for ST-segment elevation myocardial infarction. Am Heart J. 2010 Jan;159(1):55-62. doi: 10.1016/j.ahj.2009.10.033. PMID 20102867